CLINICAL TRIAL: NCT03494777
Title: Behavioral Economics Incentives to Support HIV Treatment Adherence in Sub-Saharan Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Mildmay Uganda Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH110350 (NIH); 1R01MH110350-01A1 (NIH)
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: HIV/AIDS
Keywords: ART adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two intervention arms and a control group will receive an intervention for twelve months; those not showing viral suppression at month 12 will be randomized to either continue receiving the year 1 intervention for another twelve months, or receive an additional intervention component for twelve months.
  The main analysis will be based on the sample of 330 treatment mature clients, from which the 70 treatment initiating clients will be excluded.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessor will be blinded to treatment assignment of study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adherence-based incentivization (Experimental): Participants will be eligible for prize drawings at every regular clinic visit based on high adherence as measured by MEMS-caps. In addition there will be an annual prize drawing that is conditional on showing high adherence over the course of the year.
  This arm will receive the intervention 'Incentivization based on high adherence' and the intervention 'Annual adherence prize drawing' and (if eligible) the intervention 'Year 2 booster'.
  Note: the 70 treatment initiating clients will all be assigned to this arm to receive preliminary data as to whether incentives may work for this group.
  Interventions: Behavioral: Incentivization based on high adherence; Behavioral: Annual adherence prize drawing; Behavioral: Year 2 booster
- Viral suppression-based incentivization (Experimental): Participants will be able to participate in prize drawings at every clinic visit where eligibility will be based on timely drug refills (that coincide with the clinic visits). Participants will also have a chance to enter a prize drawing at the end of every year if they show viral suppression.
  This arm will receive the intervention 'Incentivization based on timely clinic visit' and the intervention 'Annual viral suppression-based prize drawing', and (if eligible) the intervention 'Year 2 booster'.
  Interventions: Behavioral: Incentivization based on timely clinic visit; Behavioral: Annual viral suppression-based prize drawing; Behavioral: Year 2 booster
- Control (No Intervention): This arm will receive care as usual, including the adherence support mechanisms that are part of usual care practices.

INTERVENTIONS:
Behavioral: Incentivization based on high adherence — When a participant comes for a regular clinic visit, s/he will have the MEMS data extracted, and if adherence over the previous month >=90%, will participate in a prize drawing.
  Arms: Adherence-based incentivization
Behavioral: Incentivization based on timely clinic visit — When a participant comes for a regular clinic visit on the day s/he is scheduled, s/he will participate in a prize drawing.
  Arms: Viral suppression-based incentivization
Behavioral: Annual adherence prize drawing — Participants will have a chance to take part in an annual drawing where eligibility is based on the average adherence during that year.
  Arms: Adherence-based incentivization
Behavioral: Annual viral suppression-based prize drawing — Participants will have a chance to take part in an annual drawing where eligibility is based on showing viral suppression.
  Arms: Viral suppression-based incentivization
Behavioral: Year 2 booster — Those participants not showing viral suppression at month 12 will be randomized in a 1:1 fashion to receive an additional intervention component or continue receiving the same intervention arm as in Year 1.
  Arms: Adherence-based incentivization; Viral suppression-based incentivization

SUMMARY:
This study will implement an intervention in a two-year randomized controlled trial (RCT) to establish efficacy on viral suppression as a biological endpoint, compare the effectiveness of two different modes of implementation (including one entirely based on readily available clinic data), and investigate cost-effectiveness. Participants in the first intervention group (T1, n=110) will be eligible for small lottery prizes based on timely clinic visits, and qualify for an annual lottery conditional if demonstrating viral suppression; those in the second group (T2, n=110) will draw prizes conditional on electronically measured adherence at each clinic visit, and also participate in an annual lottery that is conditional on high adherence throughout the year. The control group (n=110) will receive the usual standard of care. Assessments will be conducted at baseline and then every six months. Primary outcomes are undetectable viral load and electronically measured adherence.

DETAILED DESCRIPTION:
It is imperative to find ways to boost ART adherence in sub-Saharan Africa where adherence rates have been found to decline over time, and where treatment options such as second-line regimens are limited. A promising tool is the use of incentives based on insights from behavioral economics (BE) for healthy HIV-related behavior. The proposed R01 study is based on the results of the PI's R34 'Rewarding Adherence Program (RAP)' [R34 MH096609] that demonstrated feasibility and acceptability of incentives allocated by a drawing for HIV-related behaviors, and established preliminary efficacy. The current R01 study builds on these promising results with the aim to a) use viral loads as biological endpoints that were not included in the R34 for cost reasons; b) establish efficacy in a fully powered intervention as well as comparative efficacy of two different ways of implementing the incentives including one arm that has been adapted to changing clinical guidelines and can be implemented with readily available data from clinic records; and c) assess the cost effectiveness of these two implementation modes as a further input for policy-makers. The intervention is targeted at increasing the motivation of HIV clients who have been on ART for several years through the benefit and joy of prize drawings, thereby attempting to overcome the treatment 'fatigue' that can develop in the context of mundane, daily pill taking over the course of life-long treatment. Insights from behavioral economics suggest that such an intervention may be particularly effective for people with present bias (those who have a tendency to give in to short-term temptation at the cost of more long-term benefits) that was found to be prevalent among HIV clients in the R34 study. The intervention will be implemented among 330 adult clients in three groups: for the first intervention group, timely clinic attendance will constitute the eligibility criteria for participating in a prize drawing at each scheduled clinic visit; participants are also eligible for an annual prize drawing based on showing viral suppression. The second treatment group will be incentivized on demonstrated high ART adherence between clinic visits that also determine the winning chances at an annual prize drawing. The control group will receive the usual standard of care. All participants will receive MEMS caps to record adherence and assessments over 24 months (at baseline and every 6 months thereafter). The first Specific Aim will be to evaluate the effectiveness of the intervention; the second aim is to compare the relative effectiveness of the adherence-based arm and the arm directly incentivizing viral suppression that uses only data readily available in the clinic. The third Specific Aim is to perform a comparative cost-effectiveness analysis of the two intervention arms as a further policy input. If proven efficacious, the intervention as implemented in the newly adapted arm based on viral load suppression can be readily taken over by the clinic and scaled at low cost to other clinics.

In the study also 70 treatment initiating clients (in addition to the 330 treatment mature clients described above) will be recruited, but they will be excluded from the main analysis. [Note on 9/7/2019: due to funding, we will not recruit this additional sample of treatment initiating clients]

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* at Mildmay clinic on ART for at least two years
* adherence problems in the last six months

Note: for the 70 treatment initiators to be recruited in addition to the main sample of 330 treatment-mature clients (on which the main analysis will focus), the inclusion criteria are:

* 18 years of age or older
* started on ART at Mildmay clinic within the last six months

Exclusion Criteria:

* not able to understand the consent form and study procedures
* language other than Luganda or English
* not willing to consistently use the MEMS caps device for adherence measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Electronically measured adherence | 12 months
  Number of ART doses taken / number of doses prescribed
Electronically measured adherence | 24 months
  Number of ART doses taken / number of doses prescribed
Viral suppression | At month 12
  Viral load <=200 copies/mL
Viral suppression | At month 24
  Viral load <=200 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Linnemayr, PhD, Principal Investigator — RAND
Locations (1):
- Mildmay Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wagner Z, Wang Z, Stecher C, Karamagi Y, Odiit M, Haberer JE, Linnemayr S. The association between adherence to antiretroviral therapy and viral suppression under dolutegravir-based regimens: an observational cohort study from Uganda. J Int AIDS Soc. 2024 Aug;27(8):e26350. doi: 10.1002/jia2.26350. PMID 39155425
- [Derived] Linnemayr S, Wagner Z, Saya UY, Stecher C, Lunkuse L, Wabukala P, Odiit M, Mukasa B. Behavioral Economic Incentives to Support HIV Care: Results From a Randomized Controlled Trial in Uganda. J Acquir Immune Defic Syndr. 2024 Jul 1;96(3):250-258. doi: 10.1097/QAI.0000000000003420. PMID 38534162
- [Derived] MacCarthy S, Wagner Z, Saya U, Ghai I, Karamagi Y, Odiit M, Mukasa B, Linnemayr S. Food Insecurity During the COVID-19 Pandemic: A Longitudinal Mixed-Methods Study from a Cohort of HIV Clients in Uganda. AIDS Behav. 2023 Jul;27(7):2216-2225. doi: 10.1007/s10461-022-03953-6. Epub 2023 Jan 11. PMID 36629972
- [Derived] Saya U, MacCarthy S, Mukasa B, Wabukala P, Lunkuse L, Wagner Z, Linnemayr S. "The one who doesn't take ART medication has no wealth at all and no purpose on Earth" - a qualitative assessment of how HIV-positive adults in Uganda understand the health and wealth-related benefits of ART. BMC Public Health. 2022 May 27;22(1):1056. doi: 10.1186/s12889-022-13461-w. PMID 35619119
- [Derived] MacCarthy S, Mendoza-Graf A, Jennings Mayo-Wilson L, Wagner Z, Saya U, Chemusto H, Mukasa B, Linnemayr S. A qualitative exploration of health-related present bias among HIV-positive adults in Uganda. AIDS Care. 2023 Jun;35(6):883-891. doi: 10.1080/09540121.2021.2004298. Epub 2021 Nov 21. PMID 34802344
- [Derived] Wagner Z, Mukasa B, Nakakande J, Stecher C, Saya U, Linnemayr S. Impact of the COVID-19 Pandemic on Use of HIV Care, Antiretroviral Therapy Adherence, and Viral Suppression: An Observational Cohort Study From Uganda. J Acquir Immune Defic Syndr. 2021 Dec 15;88(5):448-456. doi: 10.1097/QAI.0000000000002811. PMID 34757973
- [Derived] Jennings Mayo-Wilson L, Devoto B, Coleman J, Mukasa B, Shelton A, MacCarthy S, Saya U, Chemusto H, Linnemayr S. Habit formation in support of antiretroviral medication adherence in clinic-enrolled HIV-infected adults: a qualitative assessment using free-listing and unstructured interviewing in Kampala, Uganda. AIDS Res Ther. 2020 Jun 8;17(1):30. doi: 10.1186/s12981-020-00283-2. PMID 32513192
- [Derived] Linnemayr S, Stecher C, Saya U, MacCarthy S, Wagner Z, Jennings L, Mukasa B. Behavioral Economics Incentives to Support HIV Treatment Adherence (BEST): Protocol for a randomized controlled trial in Uganda. Trials. 2020 Jan 3;21(1):9. doi: 10.1186/s13063-019-3795-4. PMID 31900193